CLINICAL TRIAL: NCT03606200
Title: Swiss Primary Ciliary Dyskinesia Registry
Acronym: CH-PCD
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: CH-PCD (SRDR)
Record Dates: First submitted 2018-06-11; First posted 2018-07-30 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Primary Ciliary Dyskinesia; Kartagener Syndrome
MeSH Terms: conditions — Ciliary Motility Disorders; Kartagener Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 80 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Swiss Primary Ciliary Dyskinesia (PCD) Registry is a national patient registry that collects information on diagnosis, symptoms, treatment and follow-up of patients with PCD in Switzerland and provides data for national and international monitoring and research.

DETAILED DESCRIPTION:
The Swiss Primary Ciliary Dyskinesia registry (CH-PCD) was founded in 2013 as a collaborative project between epidemiologists and adult and paediatric pulmonologists. It started as a pilot project in the canton of Bern and in 2014 was extended to include all Switzerland. The data centre of the SPCDR is located at the Institute of Social and Preventive Medicine at the University of Bern. It contributes data to the international PCD registry and other international studies such as the international PCD (iPCD) cohort.

Objectives of the CH-PCD:

The Swiss Primary Ciliary Dyskinesia Registry collects information on diagnosis, symptoms, treatment and follow-up of patients with PCD in Switzerland and provides data for national and international monitoring and research. In particular, it aims to:

* Identify all patients diagnosed with PCD in Switzerland.
* Collect population based data (incidence, prevalence, time trends and regional trends).
* Document diagnostic evaluations, treatments and participation in clinical trials.
* Document the clinical course of PCD, quality of life, morbidity and mortality.
* Establish a research platform for clinical, epidemiological and basic research.

Study design:

The CH-PCD is a patient registry. At baseline (inclusion of a patient to the registry), it collects retrospectively all available data since birth and it follows included patients throughout life until death or loss to follow up, collecting prospectively data at regular time intervals.

What data is collected:

The CH-PCD collects information on demographic characteristics (e.g. age, sex), diagnostic tests and clinical data about manifestations and management of the disease. It collects repeated follow-up data on growth, lung function, clinical manifestations from all affected organ systems, microbiology and imaging, lab results, therapeutic interventions (including surgery and physiotherapy) and hospitalisations. It also collects information on neonatal symptoms related to the disease and on the symptoms, that led to referral and PCD diagnosis.

Since 2020, the CH-PCD collects through questionnaire surveys patient-reported information on symptoms and lifestyle behaviours.

Study database:

The study database is web-based, using the Research Electronic Data Capture (REDCap) platform developed at Vanderbilt University. REDCap is widely used in academic research and allows data entry and extraction in various formats.

How to participate:

Patients with PCD who would like to participate to the registry as well as physicians who treat patients with PCD should contact the CH-PCD to receive the study information and informed consent forms.

For further details, please contact: spcdr@hin.ch

Funding:

The setting up of the CH-PCD (salaries, consumables and equipment) was funded by several Swiss funding bodies, including the Lung Leagues of Bern, St. Gallen, Vaud, Ticino and Valais and the Kantonalbernischer Hilfsbund.Research activities based on data included in the CH-PCD are funded by the Swiss National Science foundation (SNF 320030_173044, 320030B_192804 and PZ00P3_185923). The CH-PCD participated to the EU funded BEAT-PCD COST Action (BM1407) and participates to the BEAT-PCD clinical research collaboration supported by the European Respiratory Society.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary ciliary dyskinesia
* Signed informed consent or assent

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages diagnosed with PCD, who are resident or treated in Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2080-12 (Estimated); Study Completion 2080-12 (Estimated)

PRIMARY OUTCOMES:
Height | every 3 months up to 80 years
  Height z-scores calculated based on available national and international references
BMI | every 3 months up to 80 years
  Body Mass Index (BMI) z-scores calculated based on available national and international references
Lung function measurements | every 3 months up to 80 years
  Spirometric indices, particularly Forced expiratory volume in 1 sec (FEV1) and Forced vital capacity (FVC) z-scores calculated based on Global Lung Function Initiative (GLI) reference values
Measurement of nasal nitric oxide using breath analyzer | at study entry (in case patient is <5 years old at study entry, then the outcome will be assessed at age 5
  Results of nasal nitric oxide measurement, performed for diagnosis
Cilia ultrastructure identified using electron microscopy analysis | at study entry
  Results of electron microscopy analysis of cilia, performed for diagnosis
Ciliary beat frequency and beat pattern using video microscopy analysis | at study entry
  Results of video microscopy analysis of cilia, performed for diagnosis
Microbiological culture of respiratory samples | every 3 months up to 80 years
  Results of microbiology cultures of respiratory samples (sputum, cough swabs, throat swabs, ear swabs, bronchoalveolar lavage) expressed in a qualitative (growth or no growth of pathogens) or semiquantitative way (the type of sample depends on the age of the patient and the clinic the sample was collected).
Antibiotic resistance of microbes isolated in microbiological cultures | every 3 months up to 80 years
  Information on antibiotic resistance of microbes isolated in microbiological cultures (see outcome 7) of respiratory samples, expressed either semiquantitatively or by the value of minimum inhibitory concentration.
Chest computed tomography | every 3 months up to 80 years
  Radiological findings from chest computed tomography
Sinus computed tomography | every 3 months up to 80 years
  Radiological findings from sinus computed tomography
Vital status | every 3 months up to 80 years
  Vital status of patient: has the patient died or is he/she still alive and in case of death what was the cause?
Clinical symptoms frequency | once a year up to 80 years
  Frequency of respiratory symptoms recorded with a patient or parent-reported questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Claudia E Kuehni, Prof, Principal Investigator — University of Bern; Myrofora Goutaki, PD, MD-PhD, Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data are shared for international collaborative projects. For requests related to IPD please contact spcdr@hin.ch

REFERENCES:
- [Result] Goutaki M, Eich MO, Halbeisen FS, Barben J, Casaulta C, Clarenbach C, Hafen G, Latzin P, Regamey N, Lazor R, Tschanz S, Zanolari M, Maurer E, Kuehni CE; Swiss PCD Registry (CH-PCD) Working Group. The Swiss Primary Ciliary Dyskinesia registry: objectives, methods and first results. Swiss Med Wkly. 2019 Jan 13;149:w20004. doi: 10.57187/smw.2019.20004. eCollection 2019 Jan 1. PMID 30691261
- [Result] Goutaki M, Husler L, Lam YT, Koppe HM, Jung A, Lazor R, Muller L; Swiss PCD Research Group; Pedersen ESL, Kuehni CE. Respiratory symptoms of Swiss people with primary ciliary dyskinesia. ERJ Open Res. 2022 Apr 11;8(2):00673-2021. doi: 10.1183/23120541.00673-2021. eCollection 2022 Apr. PMID 35415187
- [Result] Lam YT, Pedersen ESL, Schreck LD, Husler L, Koppe H, Belle FN, Clarenbach C, Latzin P; Swiss PCD research group; Kuehni CE, Goutaki M. Physical activity, respiratory physiotherapy practices, and nutrition among people with primary ciliary dyskinesia in Switzerland - a cross-sectional survey. Swiss Med Wkly. 2022 Aug 18;152:w30221. doi: 10.4414/smw.2022.w30221. eCollection 2022 Aug 15. PMID 36041191